CLINICAL TRIAL: NCT01273051
Title: CHEMORADIOTHERAPY FOR RECTAL CANCER IN THE DISTAL RECTUM FOLLOWED BY ORGANSPARING TRANSANAL ENDOSCOPIC MICROSURGERY: CARTS Study CApecitabine, Radiotherapy and Tem Surgery. A PHASE II, FEASIBILITY TRIAL
Brief Title: Transanal Endoscopic Microsurgery (TEM) After Radiochemotherapy for Rectal Cancer
Acronym: CARTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMO 2010_121
Record Dates: First submitted 2010-11-22; First posted 2011-01-10 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Rectal Tumour
Keywords: Rectal Cancer; Radiochemotherapy; TEM; Organ preservation
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Capecitabine — Capecitabine will be administered at a dose of 825 mg/m2 bid during radiotherapy treatment
Radiation: radiotherapy — radiation 25x2 Gy
Procedure: TME resection — All patients undergo a MRI of the pelvis and a rectoscopy and endorectal ultrasound 6 weeks after chemo radiation. Patients who do not respond or clinically have a T3 tumour either on visual measurements or post therapy MRI or endoanal ultrasound will be operated on with a TME resection 8 - 10 weeks after the last chemo radiation treatment.
Procedure: TEM surgery — All patients undergo a MRI of the pelvis and a rectoscopy and endorectal ultrasound 6 weeks after chemo radiation.Patients with a significant downsizing of the tumour (T0-T2) will be operated on by TEM surgery 8 -10 weeks after the last chemo radiation treatment.
  After TEM surgery, pathological assessment will dictate further treatment. Conservative treatment with careful follow-up will be performed in patients with a complete resection of a ypT0-1 rectal tumour. Patients with lymphangio invasion, an incomplete resected ypT1 (<2 mm margin), an ypT2 or ypT3 tumour after TEM will subsequently undergo TME surgery to remove the rectum within 4 weeks.

SUMMARY:
In the Netherlands approximately 2300 new patients are diagnosed with rectal cancer each year. Standard treatment for patients with a T2 or T3 rectal cancer consists of preoperative short course of radiotherapy followed by surgery. In advanced cases long course of radiotherapy combined with chemotherapy is used instead of a short cause. In some of these advanced cases a complete remission is observed after a long course of radio-/chemotherapy. Patients who respond well to neo-adjuvant treatment carry a better prognosis.

Objective of this research is to evaluate whether neo-adjuvant chemo-/radiotherapy in small non-advanced rectal cancers can be used to obtain a complete or near complete remission. In these patients could a complete resection of the rectum as an organ be avoided by treating them with a local excision with the TEM-technique (Transanal Endoscopic Microsurgery) of the scar. The advantage for these patients is, that they do not need major abdominal surgery and in a substantial number of these patients the rectum can be preserved with a better function of continence.

ELIGIBILITY:
Inclusion Criteria:

* Patients (aged >18 years) with histological proven adenocarcinoma of the distal part of the rectum (below 10 cm) without signs of distant metastases.
* T1-3 tumour without lymph nodes > 5 mm at CT, MRI and endoanal ultrasound.
* ANC > 1.5 x 109/l.
* Thrombocytes > 100 x 109/l.
* Creatinin clearance >50ml/min (according to the Cockcroft-Gault formula)
* Total serum bilirubin < 24 mol/l or below <1.5 times the upper limit of the normal.
* ASAT,ALAT: up to 5 times the upper limit.
* Colonoscopy, colonography or virtual colonoscopy should exclude synchronous colorectal lesions in other parts of the colon.
* ECOG performance score 0-2.
* Fertile women should have adequate birth control during treatment.
* Mental/physical/geographical ability to undergo treatment and follow-up.
* Written informed consent (Dutch language).

Exclusion Criteria:

* Patients with Grade 1-2 T1 tumors (can be treated with TEM surgery without chemoradiation therapy)
* Patients with circular rectal tumor or tumors who are by other means unacceptable for TEM surgery (e.g. intra anal tumors).
* Patients with faecal incontinence prior to the diagnosis of rectal cancer (complaints of soiling due to the tumor will not be an exclusion criterium).
* Severe uncontrollable medical or neurological disease.
* Patients with secondary prognosis determining malignancies.
* Patients who have been treated with radiotherapy on the pelvis.
* Use of Vitamin K antagonists.
* Fenytoine and Allopurinol use.
* Known DPD deficiency
* Uncontrolled active infection, compromised immune status, psychosis, or CNS disease.
* Pregnant or lactating women.
* Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤ 6 months prior to randomisation), myocardial infarction (≤ 6 months prior to randomisation), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication.
* Evidence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of Capecitabine or patients at high risk for treatment complications. History or evidence upon physical examination of CNS disease unless adequately treated (e.g., seizure not controlled with standard medical therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Response | Baseline and 6 weeks after chemoradiation therapy
  the response of the rectal carcinoma to chemo-/radiotherapy defined as complete response (no visible disease); partial response (more than 50% reduction of the tumour mass); no response (meaning an increase of the tumour mass less than 25% or a decrease of the tumour mass less than 50%); or progressive disease when the tumour mass increase more than 25% of the original tumour mass.

SECONDARY OUTCOMES:
Quality of life | baseline, 6-12-24 and 35 months after surgery
  Quality of life form EORTC-QLQC30 and 38. Determine the faecal continence and QOL after treatment with TEM surgery will be compared with TME treated patients.
Local Recurrence | 36 months, 60 months after surgery last enrolled patient
  Careful follow-up will determine the local recurrence rate of patients treated with TEM and TME surgery. This will be standard colorectal cancer follow-up with additional endo-anal endography and MRI for patients treated with TEM surgery during the first two years.
Toxicity | 4 weeks after surgery last enrolled patient
  Regional and systemic Toxicity/Side effects will be recorded according to the CTC-Toxicity Grading system, CTC-NCIC Toxicity Criteria v. 3.0. (See appendix to the protocol).
  Surgical and postoperative complications will be collected and assessed during interim analysis.
Number of positive lymph nodes in patient who have been treated with classical surgery | 4 weeks after surgery last enrolled patient
  The number of patients with positive lymph nodes after chemo radiation is expected to be less than 20%, this will carefully be monitored.
The number of sphincter saving procedures | 4 weeks after surgery last enrolled patient
  after organ sparing surgery by classical TEM or after TME surgery:

CONTACTS AND LOCATIONS:
Overall Officials: J.H.W de Wilt, Md PhD, Principal Investigator — University Medical Centre Nijmegen
Locations (13):
- Netherlands (13):
  - University Medical Centre Nijmegen, Nijmegen, Gelderland
  - Academisch Medisch Centrum, Amsterdam
  - NKI AVL, Amsterdam
  - Slotervaart Ziekenhuis, Amsterdam
  - Amphia Ziekenhuis, Breda
  - IJsselland Ziekenhuis, Capelle aan den IJssel
  - Catharina Ziekenhuis, Eindhoven
  - LUMC, Leiden
  - MAASTRO Clinic, Maastricht
  - Laurentius Ziekenhuis, Roermond
  - Erasmus Medical Center, Rotterdam
  - Instituut Verbeeten, Tilburg
  - Diakonessenhuis, Utrecht

REFERENCES:
- [Derived] Bokkerink GM, de Graaf EJ, Punt CJ, Nagtegaal ID, Rutten H, Nuyttens JJ, van Meerten E, Doornebosch PG, Tanis PJ, Derksen EJ, Dwarkasing RS, Marijnen CA, Cats A, Tollenaar RA, de Hingh IH, Rutten HJ, van der Schelling GP, Ten Tije AJ, Leijtens JW, Lammering G, Beets GL, Aufenacker TJ, Pronk A, Manusama ER, Hoff C, Bremers AJ, Verhoef C, de Wilt JH. The CARTS study: Chemoradiation therapy for rectal cancer in the distal rectum followed by organ-sparing transanal endoscopic microsurgery. BMC Surg. 2011 Dec 15;11:34. doi: 10.1186/1471-2482-11-34. PMID 22171697